CLINICAL TRIAL: NCT01970163
Title: A Multicenter, Randomized, Controlled, Open Label Trial of DermACELL in Subjects With Chronic Wounds of the Lower Extremities
Brief Title: DermACELL in Subjects With Chronic Wounds of the Lower Extremities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeNet Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-13-001
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic foot ulcer; Venous stasis ulcer; Wound of the lower extremity; Skin substitute; Acellular Dermal Matrix
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DermACELL (Experimental): DermACELL acellular dermal matrix will be used to treat subjects diagnosed with an ulcer of the lower extremity (diabetic foot ulcer or venous stasis ulcer).
  Interventions: Other: DermACELL
- Conventional care dressings (Placebo Comparator): Currently accepted standard of care wound management including Conventional care dressings will be utilized in subjects with a diagnosis of either diabetic foot ulcer or venous stasis ulcer.
  Interventions: Other: Conventional Care Dressings
- GraftJacket (Active Comparator): GraftJacket acellular dermal matrix will be used in those subjects diagnosed with a diabetic foot ulcer.
  Interventions: Other: GraftJacket

INTERVENTIONS:
Other: DermACELL — Acellular dermal matrix is applied at Baseline visit. The study product may be reapplied an additional time (between Weeks 2 and 12 for venous stasis ulcers and between Weeks 3 and 12 for diabetic foot ulcers).
  Other Names: LifeNet Health Product Code: DCELL112
  Arms: DermACELL
Other: GraftJacket — Acellular dermal matrix applied at Baseline visit. May be reapplied one additional time during study (between Week 2 and 12 for venous stasis ulcers and Week 3 and 12 for diabetic foot ulcers).
  Other Names: KCI Product Code: GJ44
  Arms: GraftJacket
Other: Conventional Care Dressings — Depending on the state of the wound (dry or moist), different types of nonadherent dressings would be utilized as the primary dressing:
  * If the wound is dry, a nonadherent dressing, such an oil emulsion dressing, may be appropriate, as these dressings tend to donate moisture to the wound.
  * Hydrogels can also be used if the wound is in need of moisture.
  * For a wound that is more moist, a more absorptive dressing may be more appropriate to help reduce potential for maceration.
  A secondary dressing may be desired to add either loft or cushion.
  Arms: Conventional care dressings

SUMMARY:
The study will compare treatment with DermACELL to conventional care in diabetic foot ulcers (DFU) and venous stasis ulcers (VSU).

DETAILED DESCRIPTION:
This study is designed to demonstrate the effectiveness of DermACELL in the treatment of chronic wounds of the lower extremities. DermACELL will be compared to conventional care in both subjects with diabetic foot ulcers (DFU) and subjects with venous stasis ulcers (VSU). In addition, DermACELL will be compared to an active comparator, GraftJacket, in subjects with diabetic foot ulcers.

DermACELL and GraftJacket are both made from donated human skin (dermis). These products have been processed so that cells are removed and bacteria and viruses are destroyed. This processing provided a supporting structure, an acellular dermal matrix, into which cells can migrate and divide during the wound healing process.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between the ages of 21 and 80 that are able to provide informed consent, are available for weekly clinic visits and are willing to comply with off-loading requirements of treatment;
* If diabetic, have been on a stable dose of medication to treat diabetes for less than 30 days;
* Have a DFU that has been present for at least 30 days or have a VSU that has been present for at least 60 days;

Exclusion Criteria:

* Have a DFU or VSU that is infected;
* Are pregnant or lactating;
* Have an allergy or are sensitive to one of the following antibiotics: lincomycin, gentamicin, polymyxin B, or vancomycin;
* Have a sensitivity to polysorbate 20, N-lauroyl sarcosinate, benzonase or glycerol;
* Have had a HbA1c level greater than 12% within the past 90 days;
* Have liver function tests or kidney function tests that are very elevated;
* Have a known or suspected disease of the immune system;
* Have had surgery in the past 30 days to increase blood flow into your leg or foot;
* Have cancer or a connective tissue disease (i.e. lupus, rheumatoid arthritis);
* Have undergone wound healing treatment with a living skin equivalent (i.e., Dermagraft®, Apligraf®, TheraSkin®, Oasis®, GraftJacket®, Integra®, Alloderm®) or topical growth factors in the last 4 weeks;
* Have active Charcot disease, a weakening of the bones in the foot that can occur in people who have significant nerve damage (neuropathy);

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Effect of DermACELL on the proportion of chronic wounds of the lower extremity that have healed. | 12 weeks
  The primary outcome is the comparison of the proportion of chronic wounds treated with DermACELL and treated with conventional care that have achieved 100% re-epithelialization without dressing or drainage requirements at 12 weeks. Wound closure is defined as first observation of 100% re-epithelialization without drainage or dressing requirements and complete wound closure is defined as 100% re-epithelialization without dressing or drainage requirements confirmed at two consecutive study visits 2 weeks apart.

SECONDARY OUTCOMES:
Proportion of wounds closed at 12 weeks and weekly thereafter for up to 24 weeks | 24 weeks
  The proportion of subjects with closed wounds at 12 weeks and weekly thereafter will be compared in subjects treated with DermACELL, GraftJacket (Diabetic foot ulcer subjects only) and conventional care wound management. A comparison of the proportion of subjects who received a second application of acellular dermal matrix will be made between the DermACELL and GraftJacket arms in those subjects with diabetic foot ulcers.

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events (AE), changes in vital signs, ankle-brachial index (ABI) and physical examination findings. | 24 weeks
  Safety of the interventions will be measured by the incidence of treatment-emergent AEs, changes in vital signs, ABI and physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Moore, Ph.D., Study Director — LifeNet Health, Scientific Affairs
Locations (11):
- United States (11):
  - Institute for Advanced Wound Care, Montgomery, Alabama
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - ILD Research Center, Carlsbad, California
  - Center for Clinical Research, Castro Valley, California
  - Limb Preservation Platform, Fresno, California
  - Fairfield County Foot Surgeons, Norwalk, Connecticut
  - Andrews Research and Education Institute, Gulf Breeze, Florida
  - Rosalind Franklin University, CLEAR, North Chicago, Illinois
  - Boston Medical College, Boston, Massachusetts
  - Wound Institute and Reseach Center, Dunmore, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Walters J, Cazzell S, Pham H, Vayser D, Reyzelman A. Healing Rates in a Multicenter Assessment of a Sterile, Room Temperature, Acellular Dermal Matrix Versus Conventional Care Wound Management and an Active Comparator in the Treatment of Full-Thickness Diabetic Foot Ulcers. Eplasty. 2016 Feb 4;16:e10. eCollection 2016. PMID 26933467
- [Result] Cazzell S, Vayser D, Pham H, Walters J, Reyzelman A, Samsell B, Dorsch K, Moore M. A randomized clinical trial of a human acellular dermal matrix demonstrated superior healing rates for chronic diabetic foot ulcers over conventional care and an active acellular dermal matrix comparator. Wound Repair Regen. 2017 May;25(3):483-497. doi: 10.1111/wrr.12551. Epub 2017 Jun 12. PMID 28544150